CLINICAL TRIAL: NCT06283966
Title: A Randomized, Double-blind, Parallel Group, Multi-center, Phase III Study to Assess the Efficacy of Budesonide, Glycopyrronium, and Formoterol Fumarate Metered Dose Inhaler Relative to Glycopyrronium and Formoterol Fumarate MDI on Cardiopulmonary Outcomes in Chronic Obstructive Pulmonary Disease (THARROS)
Brief Title: A Study Evaluating the Efficacy of Budesonide, Glycopyrronium and Formoterol Fumarate Metered Dosed Inhaler on Cardiopulmonary Outcomes in Chronic Obstructive Pulmonary Disease
Acronym: THARROS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5989C00001; 2023-507407-59-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: This is a Phase III randomized, double-blind, parallel group, multi-center event-driven study comparing BGF MDI 320/14.4/9.6 μg BID with GFF MDI 14.4/9.6 μg BID in participants with COPD who are at risk of a cardiopulmonary event.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BGF arm (Experimental): BGF MDI 320/14.4/9.6 μg BID
  Interventions: Drug: BGF MDI 320/14.4/9.6 μg
- GFF arm (Experimental): GFF MDI 14.4/9.6 μg BID
  Interventions: Drug: GFF MDI 14.4/9.6 μg

INTERVENTIONS:
Drug: BGF MDI 320/14.4/9.6 μg — Budesonide, glycopyrronium, and formoterol fumarate pressurized inhalation suspension
  Arms: BGF arm
Drug: GFF MDI 14.4/9.6 μg — Glycopyrronium and formoterol fumarate pressurized inhalation suspension
  Arms: GFF arm

SUMMARY:
This study will evaluate the effect of triple ICS/LAMA/LABA therapy with BGF MDI 320/14.4/9.6 μg on cardiopulmonary outcomes relative to LAMA/LABA therapy with GFF MDI 14.4/9.6 μg in a population with COPD and elevated cardiopulmonary risk.

DETAILED DESCRIPTION:
This is a Phase III randomized, double-blind, parallel group, multi-center event-driven study comparing BGF MDI 320/14.4/9.6 μg BID with GFF MDI 14.4/9.6 μg BID in participants with COPD who are at risk of a cardiopulmonary event.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants must be 40 to 80 years of age inclusive, at the time of signing

   the ICF.
2. Demonstrate acceptable MDI administration technique at Visit 1 (V1) and Visit 2 (V2)
3. A diagnosis of COPD confirmed by a post-bronchodilator FEV1/FVC ratio < 70%

   at V1.
4. Current or former smokers with a history of at least 10 pack-years of cigarette smoking;

   defined as (number of cigarettes per day/20) x number of years smoked. Previous smokers are defined as those who have stopped smoking for at least 6

   months prior to V1.
5. A baseline peripheral blood eosinophil count of ≥ 100 cells/mm3 assessed at Visit 1 by

   the central laboratory
6. A CAT score of ≥ 10 at Visit 1.
7. Participant must fulfill at least 1 of the 4 CV disease/risk factor criteria below [(a), (b),

   (c), or (d)]:
   1. : Established CV Disease
   2. : Combination of CV risk factors:

      * Hypertension
      * Diabetes Mellitus
      * Chronic Kidney Disease
      * Dyslipidemia
      * Obesity
   3. : High risk of CV disease determined using an established CV risk assessment

      tool.
   4. : CT coronary Artery Calcification
8. Willing and, in the opinion of the investigator, able to adjust current COPD therapy, as

   required by the protocol.
9. Willing to visit at the study site or participate in virtual visits as required per the protocol

   to complete all study assessments.
10. A female is eligible to enter and participate in the study if the female is of:

    * Non-childbearing potential: either permanently sterilized or who are post-menopausal.
    * Childbearing potential: has a negative serum pregnancy test at V1 and must use one

    highly effective form of birth control.
11. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in the protocol.

Exclusion Criteria:

1. Active diagnosis of asthma within the past 5 years (previous diagnosis as a child or adolescent are eligible), asthma-COPD overlap, or any other chronic respiratory disease other than COPD such as alpha-1 antitrypsin deficiency, active tuberculosis, lung fibrosis, sarcoidosis, interstitial lung disease, and pulmonary hypertension.
2. End-stage renal disease requiring renal replacement therapy
3. History of heart or lung transplant or actively listed for heart or lung transplant.
4. Implanted left ventricular assist device or implant anticipated in < 3 months.
5. History of lung cancer and/or treatment for lung cancer within the 5 years prior to Visit 1.
6. Unstable or life-threatening cardiac disease - participants with any of the following at Visit 1 would be excluded:

   1. An MI or unstable angina in the last 8 weeks
   2. Unstable or life-threatening cardiac arrhythmia requiring intervention in the last 8 weeks.

   NOTE: Any participant who experiences unstable or life-threatening cardiac disease during the run-in period will be excluded but can be rescreened 8 weeks after the resolution of the event.
7. Pneumonia and/or moderate or severe COPD exacerbation that has not resolved at least 8 weeks prior to Visit 1
8. Any life-threatening condition, including malignancy, with a life expectancy < 5 years, other than CV disease or COPD, that might prevent the participant from completing the study.
9. Use of maintenance ICS treatment within the past 12 months.
10. Unable to abstain from protocol-defined prohibited medications
11. Participation in another clinical study with a study intervention administered in the last 30 days or 5 half-lives, whichever is longer prior to Visit 1 (any other investigational product that is not identified in protocol is prohibited for use during the duration of the study).
12. Participants with a known hypersensitivity to LAMA, LABA or ICS or any component of the MDI.
13. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
14. Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.
15. Previous randomization in the present study.
16. For females only - currently pregnant (confirmed with positive pregnancy test) or breastfeeding

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2028-03-07 (Estimated); Study Completion 2028-03-07 (Estimated)

PRIMARY OUTCOMES:
Time to first severe cardiac or COPD event | Up to 3 years
  Evaluate the effect of combination triple therapy (BGF MDI 320/14.4/9.6 μg) compared with dual bronchodilator therapy (GFF MDI 14.4/9.6 μg) on cardiopulmonary outcomes.

SECONDARY OUTCOMES:
Time to first severe COPD exacerbation event | Up to 3 years
  Evaluate the effect of combination triple therapy (BGF MDI 320/14.4/9.6 μg) compared with dual bronchodilator therapy (GFF MDI 14.4/9.6 μg) on severe COPD exacerbations.
Time to first severe cardiac event | Up to 3 years
  Evaluate the effect of combination triple therapy (BGF MDI 320/14.4/9.6 μg) compared with dual bronchodilator therapy (GFF MDI 14.4/9.6 μg) on severe cardiac outcomes.
Time to cardiopulmonary death | Up to 3 years
  Evaluate the effect of combination triple therapy (BGF MDI 320/14.4/9.6 μg) compared with dual bronchodilator therapy (GFF MDI 14.4/9.6 μg) on cardiopulmonary deaths.
Moderate/severe COPD exacerbation rate | Over time, up 3 years
  Evaluate the effect of combination triple therapy (BGF MDI 320/14.4/9.6 μg) compared with dual bronchodilator therapy (GFF MDI 14.4/9.6 μg) on moderate/severe COPD exacerbations.
Time to Myocardial Infarction (MI) hospitalization or cardiac death | Up to 3 years
  Evaluate the effect of combination triple therapy (BGF MDI 320/14.4/9.6 μg) compared with dual bronchodilator therapy (GFF MDI 14.4/9.6 μg) on the time to MI hospitalization (or cardiac death).
Time to Heart Failure (HF) acute healthcare visit/hospitalization or cardiac death | Up to 3 years
  Evaluate the effect of combination triple therapy (BGF MDI 320/14.4/9.6 μg) compared with dual bronchodilator therapy (GFF MDI 14.4/9.6 μg) on the time to HF acute healthcare visit/hospitalization (or cardiac death).

OTHER OUTCOMES:
Serious Adverse Events (SAEs) and Adverse Events leading to discontinuation (DAEs), Adverse Events of Special Interest (AESIs) of pneumonia leading to hospitalization or death | Up to 3 years
  To assess the safety and tolerability of BGF MDI and GFF MDI

CONTACTS AND LOCATIONS:
Locations (701):
- United States (191):
  - Research Site, Athens, Alabama
  - Research Site, Cullman, Alabama
  - Research Site, Fairhope, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Sheffield, Alabama
  - Research Site, Gilbert, Arizona
  - Research Site, Glendale, Arizona
  - Research Site, Mesa, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tempe, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Apple Valley, California
  - Research Site, Canoga Park, California
  - Research Site, Castroville, California
  - Research Site, Garden Grove, California
  - Research Site, Gardena, California
  - Research Site, Inglewood, California
  - Research Site, La Mesa, California
  - Research Site, La Palma, California
  - Research Site, Lomita, California
  - Research Site, Long Beach, California
  - Research Site, Los Alamitos, California
  - Research Site, Newport Beach, California
  - Research Site, North Hollywood, California
  - Research Site, Pomona, California
  - Research Site, Sacramento, California
  - Research Site, San Bernardino, California
  - Research Site, San Diego, California
  - Research Site, San Dimas, California
  - Research Site, Santa Ana, California
  - Research Site, Tarzana, California
  - Research Site, Thousand Oaks, California
  - Research Site, Van Nuys, California
  - Research Site, Vista, California
  - Research Site, Westminster, California
  - Research Site, Aurora, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Englewood, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Boynton Beach, Florida
  - Research Site, Bradenton, Florida
  - Research Site, Cape Coral, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Crystal River, Florida
  - Research Site, Cutler Bay, Florida
  - Research Site, Edgewater, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Homestead, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Lake City, Florida
  - Research Site, Lake Worth, Florida
  - Research Site, Lakeland, Florida
  - Research Site, Loxahatchee Groves, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Naples, Florida
  - Research Site, Ocala, Florida
  - Research Site, Orlando, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Plantation, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Sun City Center, Florida
  - Research Site, Tamarac, Florida
  - Research Site, Tampa, Florida
  - Research Site, Fayetteville, Georgia
  - Research Site, Peachtree Corners, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Tucker, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Winfield, Illinois
  - Research Site, Valparaiso, Indiana
  - Research Site, Sioux City, Iowa
  - Research Site, Newton, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Paducah, Kentucky
  - Research Site, Lafayette, Louisiana
  - Research Site, Monroe, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Zachary, Louisiana
  - Research Site, Glen Burnie, Maryland
  - Research Site, Oxon Hill, Maryland
  - Research Site, Potomac, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Flint, Michigan
  - Research Site, Southfield, Michigan
  - Research Site, Gulfport, Mississippi
  - Research Site, Olive Branch, Mississippi
  - Research Site, Kansas City, Missouri
  - Research Site, Liberty, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Missoula, Montana
  - Research Site, Fremont, Nebraska
  - Research Site, Grand Island, Nebraska
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Lawrence, New Jersey
  - Research Site, Mullica Hill, New Jersey
  - Research Site, Toms River, New Jersey
  - Research Site, Union City, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Albany, New York
  - Research Site, Bronxville, New York
  - Research Site, Brooklyn, New York
  - Research Site, Massapequa, New York
  - Research Site, New Windsor, New York
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Vestal, New York
  - Research Site, Fayetteville, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Huntersville, North Carolina
  - Research Site, Morehead City, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Salisbury, North Carolina
  - Research Site, Statesville, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Beavercreek, Ohio
  - Research Site, Blue Ash, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Marion, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Norman, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Grants Pass, Oregon
  - Research Site, Medford, Oregon
  - Research Site, Roseburg, Oregon
  - Research Site, Camp Hill, Pennsylvania
  - Research Site, DuBois, Pennsylvania
  - Research Site, Exton, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Anderson, South Carolina
  - Research Site, Charleston, South Carolina
  - Research Site, Columbia, South Carolina
  - Research Site, Gaffney, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Union, South Carolina
  - Research Site, Pierre, South Dakota
  - Research Site, Rapid City, South Dakota
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Chattanooga, Tennessee
  - Research Site, Elizabethton, Tennessee
  - Research Site, Franklin, Tennessee
  - Research Site, Morristown, Tennessee
  - Research Site, Tullahoma, Tennessee
  - Research Site, Abilene, Texas
  - Research Site, Amarillo, Texas
  - Research Site, Austin, Texas
  - Research Site, Brownsville, Texas
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Forney, Texas
  - Research Site, Georgetown, Texas
  - Research Site, Houston, Texas
  - Research Site, Katy, Texas
  - Research Site, Kerrville, Texas
  - Research Site, Kingwood, Texas
  - Research Site, Lewisville, Texas
  - Research Site, McAllen, Texas
  - Research Site, McKinney, Texas
  - Research Site, Paris, Texas
  - Research Site, Plano, Texas
  - Research Site, Victoria, Texas
  - Research Site, Waco, Texas
  - Research Site, Wichita Falls, Texas
  - Research Site, Wylie, Texas
  - Research Site, Bountiful, Utah
  - Research Site, Ogden, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, West Jordan, Utah
  - Research Site, West Valley City, Utah
  - Research Site, Newport News, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Suffolk, Virginia
  - Research Site, Spokane, Washington
  - Research Site, Morgantown, West Virginia
  - Research Site, Cudahy, Wisconsin
  - Research Site, Milwaukee, Wisconsin
- Argentina (12):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Capital Federal
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Florida
  - Research Site, Mar del Plata
  - Research Site, Mendoza
  - Research Site, Ranelagh
  - Research Site, Rosario
  - Research Site, San Fernando
  - Research Site, San Juan Bautista
  - Research Site, San Miguel de Tucumán
- Australia (11):
  - Research Site, Birtinya
  - Research Site, Cairns
  - Research Site, Chermside
  - Research Site, Coffs Harbour
  - Research Site, Dubbo
  - Research Site, Nedlands
  - Research Site, Port Macquarie
  - Research Site, Spearwood
  - Research Site, St Albans
  - Research Site, Waitara
  - Research Site, Wangaratta
- Austria (5):
  - Research Site, Bad Ischl
  - Research Site, Braunau am Inn
  - Research Site, Feldbach
  - Research Site, Graz
  - Research Site, Vienna
- Brazil (26):
  - Research Site, Belo Horizonte
  - Research Site, Blumenau
  - Research Site, Brasília
  - Research Site, Campina Grande do Sul
  - Research Site, Campinas
  - Research Site, Caxias do Sul
  - Research Site, Curitiba
  - Research Site, Fortaleza
  - Research Site, Ijuí
  - Research Site, Juiz de Fora
  - Research Site, Mossoró
  - Research Site, Natal
  - Research Site, Niterói
  - Research Site, Passo Fundo
  - Research Site, Porto Alegre
  - Research Site, Recife
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, Santo André
  - Research Site, São Bernardo do Campo
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
  - Research Site, Serra
  - Research Site, Sorocaba
  - Research Site, Volta Redonda
  - Research Site, Votuporanga
- Bulgaria (21):
  - Research Site, Burgas
  - Research Site, Dobrich
  - Research Site, Dupnitsa
  - Research Site, Haskovo
  - Research Site, Kozloduy
  - Research Site, Montana
  - Research Site, Panagyurishte
  - Research Site, Pazardzhik
  - Research Site, Pernik
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sandanski
  - Research Site, Sevlievo
  - Research Site, Sliven
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Varna
  - Research Site, Vidin
  - Research Site, Vratsa
  - Research Site, Yambol
- Canada (17):
  - Research Site, Calgary, Alberta
  - Research Site, Sherwood Park, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, Richmond, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Sydney, Nova Scotia
  - Research Site, Ajax, Ontario
  - Research Site, Guelph, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Thunder Bay, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Trois-Rivières, Quebec
  - Research Site, Saskatoon, Saskatchewan
- Chile (8):
  - Research Site, Curicó
  - Research Site, Quillota
  - Research Site, Santiago
  - Research Site, Talca
  - Research Site, Temuco
  - Research Site, Victoria
  - Research Site, Viña del Mar
  - Research Site, Vitacura
- China (68):
  - Research Site, Anning
  - Research Site, Anyang
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Changzhi
  - Research Site, Chengdu
  - Research Site, Chifeng
  - Research Site, Chizhou
  - Research Site, Chongqing
  - Research Site, Daqing
  - Research Site, Dazhou
  - Research Site, Foshan
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Heze
  - Research Site, Hohhot
  - Research Site, Huizhou
  - Research Site, Jiaozuo
  - Research Site, Jinhua
  - Research Site, Jining
  - Research Site, Kaifeng
  - Research Site, Langfang
  - Research Site, Lanzhou
  - Research Site, Lishui
  - Research Site, Liuchow
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanyang
  - Research Site, Pingxiang
  - Research Site, Qingdao
  - Research Site, Qingyuan
  - Research Site, Ruian
  - Research Site, Sanya
  - Research Site, Shanghai
  - Research Site, Shantou
  - Research Site, Shaoxing
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Shihezi
  - Research Site, Shijiazhuang
  - Research Site, Siping
  - Research Site, Suining Shi
  - Research Site, Taicang
  - Research Site, Taiyuan
  - Research Site, Taizhou
  - Research Site, Ürümqi
  - Research Site, Weifang
  - Research Site, Wenzhou
  - Research Site, Xi'an
  - Research Site, Xiamen
  - Research Site, Xiangtan
  - Research Site, Xianyang
  - Research Site, Xingtai
  - Research Site, Xinxiang
  - Research Site, Xuzhou
  - Research Site, Yangzhou
  - Research Site, Yinchuan
  - Research Site, Zaozhuang
  - Research Site, Zhangzhou
  - Research Site, Zhengzhou
  - Research Site, Zhuhai
  - Research Site, Zhumadian
  - Research Site, Zhuzhou
  - Research Site, Zigong
- Colombia (7):
  - Research Site, Armenia
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Manizales
  - Research Site, Medellín
  - Research Site, Piedecuesta
  - Research Site, Rionegro
- Czechia (7):
  - Research Site, Brandýs nad Labem
  - Research Site, Jindřichův Hradec
  - Research Site, Olomouc
  - Research Site, Ostrava
  - Research Site, Prague
  - Research Site, Rokycany
  - Research Site, Tábor
- Denmark (6):
  - Research Site, Aalborg
  - Research Site, Esbjerg
  - Research Site, Hvidovre
  - Research Site, København NV
  - Research Site, Næstved
  - Research Site, Vejle
- Finland (4):
  - Research Site, Helsinki
  - Research Site, Kangasala
  - Research Site, Kuopio
  - Research Site, Turku
- France (26):
  - Research Site, Aix-en-Provence
  - Research Site, Aurillac
  - Research Site, Bayonne
  - Research Site, Biarritz
  - Research Site, Blois
  - Research Site, Brest
  - Research Site, Cannes
  - Research Site, Cherbourg
  - Research Site, Créteil
  - Research Site, La Tronche
  - Research Site, Laval
  - Research Site, Le Coudray
  - Research Site, Lomme
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Mulhouse
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Pringy
  - Research Site, Quint-Fonsegrives
  - Research Site, Reims
  - Research Site, Roscoff
  - Research Site, Strasbourg
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Vannes
  - Research Site, Villeurbanne
- Germany (36):
  - Research Site, Ahrensburg
  - Research Site, Augsburg
  - Research Site, Bamberg
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Bremen
  - Research Site, Cottbus
  - Research Site, Dachau
  - Research Site, Darmstadt
  - Research Site, Deggingen
  - Research Site, Dresden
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Ibbenbueren
  - Research Site, Karlsruhe
  - Research Site, Landsberg
  - Research Site, Leipzig
  - Research Site, Lübeck
  - Research Site, Mainz
  - Research Site, Marburg
  - Research Site, Moers
  - Research Site, München
  - Research Site, Offenbach
  - Research Site, Peine
  - Research Site, Rheine
  - Research Site, Riesa
  - Research Site, Rosenheim
  - Research Site, Solingen
  - Research Site, Wallerfing
  - Research Site, Weißenburg
  - Research Site, Wermsdorf
  - Research Site, Wiesbaden
  - Research Site, Witten
- Greece (4):
  - Research Site, Athens
  - Research Site, Ioannina
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Hungary (21):
  - Research Site, Balatonfüred
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Edelény
  - Research Site, Encs
  - Research Site, Gödöllő
  - Research Site, Gyöngyös - Mátraháza
  - Research Site, Hajdúnánás
  - Research Site, Kalocsa
  - Research Site, Komádi
  - Research Site, Monor
  - Research Site, Pécs
  - Research Site, Püspökladány
  - Research Site, Százhalombatta
  - Research Site, Szeged
  - Research Site, Székesfehérvár
  - Research Site, Szolnok
  - Research Site, Tapolca
  - Research Site, Törökbálint
  - Research Site, Vajszló
- India (17):
  - Research Site, Ahmedabad
  - Research Site, Aligarh
  - Research Site, Belagavi
  - Research Site, Calicut
  - Research Site, Chandigarh
  - Research Site, Dehradun
  - Research Site, Delhi
  - Research Site, Dwārka
  - Research Site, Hyderabad
  - Research Site, Jaipur
  - Research Site, Kolkata
  - Research Site, Mangalore
  - Research Site, Mumbai
  - Research Site, Nagpur
  - Research Site, New Delhi
  - Research Site, Pune
  - Research Site, Vijayawada
- Italy (12):
  - Research Site, Ancona
  - Research Site, Florence
  - Research Site, Genoa
  - Research Site, Mestre
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Pavia
  - Research Site, Perugia
  - Research Site, Roma
  - Research Site, Rome
  - Research Site, Siena
  - Research Site, Varese
- Japan (18):
  - Research Site, Chūōku
  - Research Site, Fujieda-shi
  - Research Site, Fukuoka
  - Research Site, Kitakyushu
  - Research Site, Kobe
  - Research Site, Kure-shi
  - Research Site, Kyoto
  - Research Site, Minoh
  - Research Site, Mizunami-shi
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Osaki-shi
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
  - Research Site, Takamatsu
  - Research Site, Yamagata
  - Research Site, Yanagawa-shi
  - Research Site, Yokohama
- Malaysia (8):
  - Research Site, Alor Star
  - Research Site, Kajang
  - Research Site, Kuala Lumpur
  - Research Site, Kuala Pilah
  - Research Site, Sandakan
  - Research Site, Sarawak Miri
  - Research Site, Seremban
  - Research Site, Sibu
- Mexico (15):
  - Research Site, Benito Juárez
  - Research Site, Chihuahua City
  - Research Site, Cuernavaca
  - Research Site, Culiacán
  - Research Site, Guadalajara
  - Research Site, Juriquilla
  - Research Site, Metepec
  - Research Site, Mexico City
  - Research Site, Mérida
  - Research Site, Monterrey
  - Research Site, Oaxaca City
  - Research Site, Tijuana
  - Research Site, Veracruz
  - Research Site, Xalapa
  - Research Site, Zapopan
- Norway (4):
  - Research Site, Kongsberg
  - Research Site, Lørenskog
  - Research Site, Skedsmokorset
  - Research Site, Trondheim
- Peru (3):
  - Research Site, El Agustino
  - Research Site, Lima
  - Research Site, Piura
- Philippines (11):
  - Research Site, Dagupan
  - Research Site, Iloilo City
  - Research Site, Las Piñas
  - Research Site, Mabalacat
  - Research Site, Manadaluyong City
  - Research Site, Manila
  - Research Site, Marilao
  - Research Site, Puerto Princesa City
  - Research Site, Quezon City
  - Research Site, Roxas City
  - Research Site, Tondo
- Poland (29):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Chęciny
  - Research Site, Chojnice
  - Research Site, Częstochowa
  - Research Site, Inowrocław
  - Research Site, Karczew
  - Research Site, Katowice
  - Research Site, Kielce
  - Research Site, Krakow
  - Research Site, Libiąż
  - Research Site, Lodz
  - Research Site, Lubin
  - Research Site, Lublin
  - Research Site, Ostrowiec Świętokrzyski
  - Research Site, Piaseczno
  - Research Site, Poznan
  - Research Site, Płock
  - Research Site, Rzeszów
  - Research Site, Sieradz
  - Research Site, Skórzewo
  - Research Site, Sochaczew
  - Research Site, Sosnowiec
  - Research Site, Szczecin
  - Research Site, Słupsk
  - Research Site, Torun
  - Research Site, Ustroń
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Romania (7):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Leamna de Sus
  - Research Site, Negreşti-Oaş
  - Research Site, Oradea
  - Research Site, Târgu Mureş
  - Research Site, Timișoara
- Serbia (5):
  - Research Site, Belgrade
  - Research Site, Kamenitz
  - Research Site, Kragujevac
  - Research Site, Niš
  - Research Site, Novi Sad
- Slovakia (8):
  - Research Site, Bratislava
  - Research Site, Brezno
  - Research Site, Humenné
  - Research Site, Košice
  - Research Site, Kráľovský Chlmec
  - Research Site, Levice
  - Research Site, Prešov
  - Research Site, Topoľčany
- South Korea (8):
  - Research Site, Anyang-si
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Gwangju
  - Research Site, Jeonju
  - Research Site, Seoul
  - Research Site, Uijeongbu-si
  - Research Site, Ulsan
- Spain (15):
  - Research Site, Alicante
  - Research Site, Badia Del Vallès
  - Research Site, Barakaldo
  - Research Site, Barcelona
  - Research Site, Castro Urdiales
  - Research Site, Córdoba
  - Research Site, Granada
  - Research Site, Madrid
  - Research Site, Marbella (Málaga)
  - Research Site, Mataró
  - Research Site, Málaga
  - Research Site, Palma
  - Research Site, Patraix
  - Research Site, Santa Cruz de Tenerife
  - Research Site, Santiago de Compostela-Coruña
- Sweden (9):
  - Research Site, Danderyd
  - Research Site, Gothenburg
  - Research Site, Höllviken
  - Research Site, Kungsbacka
  - Research Site, Lund
  - Research Site, Örebro
  - Research Site, Stockholm
  - Research Site, Umeå
  - Research Site, Uppsala
- Taiwan (8):
  - Research Site, Changhua County
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan
  - Research Site, Taoyuan District
  - Research Site, Yunlin
- Thailand (8):
  - Research Site, Bang Kra So
  - Research Site, Bangkok
  - Research Site, Hat Yai
  - Research Site, Khlong Luang
  - Research Site, Muang
  - Research Site, Ongkharak
  - Research Site, Phitsanulok
  - Research Site, Ratchathewi
- Turkey (Türkiye) (14):
  - Research Site, Adana
  - Research Site, Afyonkarahisar
  - Research Site, Antalya
  - Research Site, Bursa
  - Research Site, Çanakkale
  - Research Site, Çankaya
  - Research Site, Isparta
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kayseri
  - Research Site, Kocaeli
  - Research Site, Mersin
  - Research Site, Tekirdağ
  - Research Site, Zeytinburnu
- Ukraine (8):
  - Research Site, Chernivtsi
  - Research Site, Chernivtsі
  - Research Site, Ivano-Frankivsk
  - Research Site, Kyiv
  - Research Site, Lviv
  - Research Site, Ternopil
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
- United Kingdom (24):
  - Research Site, Bicester
  - Research Site, Bollington
  - Research Site, Bradford
  - Research Site, Cardiff
  - Research Site, Chesterfield
  - Research Site, Corby
  - Research Site, Cottingham
  - Research Site, Fowey
  - Research Site, Glasgow
  - Research Site, Hounslow
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newquay
  - Research Site, North Somerset
  - Research Site, Northallerton
  - Research Site, Norwich
  - Research Site, Nottingham
  - Research Site, Perth
  - Research Site, Poole
  - Research Site, Sheffield
  - Research Site, Torbay
  - Research Site, Whitney
  - Research Site, Witney

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home